CLINICAL TRIAL: NCT05716711
Title: The Effect of Different Essential Oils in Stoma Bags on Deodorization, Life Satisfaction, Stoma Adaptation in Individuals With Colostomy
Brief Title: Essential Oils in Stoma Bags on Deodorization, Life Satisfaction, Stoma Adaptation in Individuals With Colostomy
Acronym: surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, dudu alptekin, PHD STUDENT, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: rid27463
Record Dates: First submitted 2022-07-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Stoma Site Odor
Keywords: COLOSTOMY, ODOR, LIFE SATISFACTION, STOMA HARMONY,
MeSH Terms: conditions — Personal Satisfaction | interventions — lavender oil; SPEN protein, human

STUDY DESIGN:
Intervention Model Description: GROUP 1 GROUP2 CONTROL GROUP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (Experimental): GROUP 1
  1st GROUP LAVENDER OIL EXTRACT WILL BE APPLIED TO 20 PATIENTS WITH COLOSTOMY FOR 1 MONTH WITH 20 DROPS A DAY INTO THE STOMA BAG
  Interventions: Other: LAVENDER OIL
- GROUP 2 (Experimental): 2nd GROUP MINT OIL EXTRACT WILL BE APPLIED TO 20 PATIENTS WITH COLOSTOMY DURING 1 MONTH.
  Interventions: Other: LAVENDER OIL
- CONTROL GROUP (No Intervention): 20 PATIENTS WITH COLOSTOMY WITH NO INTERVENTION

INTERVENTIONS:
Other: LAVENDER OIL — IT WILL BE APPLIED TO 60 PATIENTS, 20 IN EACH GROUP, WITH A COLOSTOMY
  Other Names: MINT OIL; NON-INTERVENTION
  Arms: GROUP 1; GROUP 2

SUMMARY:
This study was planned to examine the effects of using the lavender essential oil and peppermint essential oil in stoma bags on odor removal, life satisfaction, and stoma compliance in patients with a stoma.

DETAILED DESCRIPTION:
There are commercially available products that health insurance does not pay for to eliminate the odor caused by gas and stool output in patients with colostomy. The limited variety of these products in our country makes it difficult for patients to access the product. In addition, it was seen in the patient feedback that they thought these products had chemical content and were worried that they would damage the colostomy. For these reasons, there was a need to search for more accessible, affordable, and non-chemical products. Essential oils are volatile, aromatic, concentrated oily liquids taken from the essence of various plant parts. Research results on the antibacterial, antifungal, antiviral, antioxidative, and antimutagenic effects of plant essential oils are generally positive. Lavender essential oil and peppermint essential oil have been used in the past, for reasons such as creating a pleasant smell, providing wound healing, antibacterial and anxiolytic properties, and improving the quality of life. For this reason, it is accepted that the use of herbal essential oil and extract can be one effective solution. In the study of Kazemi et al. (2021); Lavender essential oil has also been found to be effective in wound healing. In Duluklu's (2018) study on patients with colostomy, it was determined that there was a significant improvement in the living conditions of the experimental group formed by dripping lavender oil into the colostomy bag. It was observed that there was a significant difference between the stoma compliance scale acceptance sub-dimension and the overall stoma compliance mean score. In rainbow trout, Metin et al. (2015), in his study; They found that the use of peppermint oil did not cause any toxic effects on fish. Anderson et al.) in a randomized double-blind study with individuals experiencing postoperative nausea and vomiting, given lisinopril alcohol, peppermint oil, and placebo (saline) effective products, and nausea determined at the second and fifth minutes following inhalation of peppermint oil applied to gauze before the application of peppermint oil extract. It was determined that it decreased significantly according to the feeling of nausea. In literature reviews; There are limited studies on using lavender essential oil for odor removal in individuals with colostomy. There is no use of peppermint essential oil. Using lavender oil and peppermint oil in a stoma bag is a simple, natural, and low-cost method for odor removal.

ELIGIBILITY:
Inclusion Criteria:

* Have a stoma
* To be compatible with essential oils

Exclusion Criteria:

* Patients with allergic reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
The Effect of Different Essential Oils in Stoma Bags on Deodorization, Life Satisfaction, Stoma Adaptation in Individuals with Colostomy | 1 month
  İn patients with a permanent stoma; The level of discomfort from odor was measured by a questionnaire study using a numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: dudu alptekin, Principal Investigator — Cukurova University
Locations (1):
- Çukurova Üniversitesi, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
BETWEEN 2020 - 2022
Supporting Information: Study Protocol, SAP
Time Frame: 2020-2022
Access Criteria: FROM THE PATIENTS APPLYING TO THE STOMATHERAPY UNIT PATIENTS MEETING THE WORKING CRITERIA

REFERENCES:
- [Derived] Alptekin D, Arslan S. The effect of different essential oils used in stoma bags of individuals with colostomy remooval of odor, life satisfaction and effect on stoma fit: Randomized controlled study. Explore (NY). 2024 Nov-Dec;20(6):103065. doi: 10.1016/j.explore.2024.103065. Epub 2024 Oct 9. PMID 39418824